CLINICAL TRIAL: NCT00101543
Title: Gait Training For Acute Stroke: FNS and Weight Supported Treadmill Training
Brief Title: Gait Training For Acute Stroke: Functional Neuromuscular Stimulation (FNS) and Weight Supported Treadmill Training
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A3102R
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2005-01

CONDITIONS: Stroke
Keywords: Gait Training; Motor learning; Electrical stimulation; Body Weight supported Treadmill Training; Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Electric Stimulation

INTERVENTIONS:
Device: Electrical Stimulation with Intramuscular Electrodes
Procedure: Body Weight Supported Treadmill Training

SUMMARY:
Conventional rehabilitation does not restore normal, safe gait to many stroke survivors. Functional neuromuscular stimulation (FNS) using intramuscular (IM) electrodes (FNS-IM) improved persistent gait deficits for patients with chronic stroke (1-7 years post stroke), but required a long protocol of 6-18 months. For chronic deficits, a shortened response to treatment (3 months) was obtained by combining FNS-IM with body weight-supported treadmill training (BWSTT). Gains included strength, coordination, gait kinematics, walking endurance, and quality of life. Gait deficits treated in the chronic phase are more resistant to treatment than in the early recovery phase, because chronic, abnormal movement patterns are more ingrained. Therefore, during the early recovery phase, it is likely that a relatively greater treatment response will be obtained. The purpose of the proposed work is to test the combination FNS-IM + BWSTT during the early recovery phase following stroke. Hypothesis I is: FNS-IM + BWSTT will restore volitional gait more completely for subjects during the early recovery phase following stroke, compared to BWSTT alone. Subjects will be admitted at 1-11 months after stroke. Thirty five subjects will be randomized to one of the two treatment groups. They will be treated for 48 sessions, four sessions/week. Primary outcome measures will be: kinematic swing phase gait components, energy cost of gait, and an index of walking endurance. Secondary outcome measures will be kinematic stance phase gait components and gait speed. The second set of hypotheses will test the relationship between restoration of mobility and measurements of impairment, function and quality of life.

DETAILED DESCRIPTION:
Conventional rehabilitation does not restore normal, safe gait to many stroke survivors. Functional neuromuscular stimulation (FNS) using intramuscular (IM) electrodes (FNS-IM) improved persistent gait deficits for patients with chronic stroke (1-7 years post stroke), but required a long protocol of 6-18 months. For chronic deficits, a shortened response to treatment (3 months) was obtained by combining FNS-IM with body weight-supported treadmill training (BWSTT). Gains included strength, coordination, gait kinematics, walking endurance, and quality of life. Gait deficits treated in the chronic phase are more resistant to treatment than in the early recovery phase, because chronic, abnormal movement patterns are more ingrained. Therefore, during the early recovery phase, it is likely that a relatively greater treatment response will be obtained. The purpose of the proposed work is to test the combination FNS-IM + BWSTT during the early recovery phase following stroke. Hypothesis I is: FNS-IM + BWSTT will restore volitional gait more completely for subjects during the early recovery phase following stroke, compared to BWSTT alone. Subjects will be admitted at 1-11 months after stroke. Thirty five subjects will be randomized to one of the two treatment groups. They will be treated for 48 sessions, four sessions/week. Primary outcome measures will be: kinematic swing phase gait components, energy cost of gait, and an index of walking endurance. Secondary outcome measures will be kinematic stance phase gait components and gait speed. The second set of hypotheses will test the relationship between restoration of mobility and measurements of impairment, function and quality of life. Additionally, co-variates will be assessed at entry into the study: gender, age, mood, co-morbidities, time since stroke, and weeks of prior rehabilitation. Data for outcome measures will be collected at weeks 1, 6, 12, and 6 months after the end of treatment. For Hypothesis I testing, contrasts will be made between the two treatment groups. A separate regression model will be analyzed for each outcome measure. The post-test score for a given primary outcome measure will serve as the dependent variable in a regression model. The two independent variables will be the treatment assignment information (as a dichotomous variable) and the pretest score on the given outcome measure (the covariate). In additional model analyses for the second set of hypotheses, the relationships will be ascertained between mobility restoration and impairment, function, and quality of life. Mobility deficits following stroke pose a significant economic, social, and psychological hardship to the individual and to society. Development of techniques that improve lower extremity function will improve the quality of life and reduce associated health care costs for patients after stroke. The results of the proposed study have the potential to provide a new acute stroke treatment that will increase the rate of recovery, produce a more comprehensive recovery of motor function, safer gait, greater functional independence, and enhanced quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Stroke 1-11 months ago
* Inability to move leg normally

Exclusion Criteria:

* Pacemaker
* Progressive medical condition (i.e. Parkinsons Disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2003-08; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland VA Medical Center; Research Service, Cleveland, Ohio, United States